CLINICAL TRIAL: NCT01729273
Title: Vascular Health and Exercise Performance of Overweight Children in 12 Weeks Using Skype
Brief Title: Vascular Health and Exercise Performance of Overweight Children
Acronym: VHEPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHRI-23724
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diet and Exercise Intervention (Experimental): Tests will include EndoPAT analysis to assess endothelial function, applanation tonometry to assess arterial stiffness, carotid artery imaging to assess the wall thickness of the carotid arteries, exercise testing to assess the physical exercise capacity of these children and blood work to evaluate the lipid profile and inflammation status (CRP).
  The Home Exercise Program will be 3 days a week for 12 weeks and participants will connect with the trainer to perform 45-60 minutes of a combination of strength training and aerobic activity via Skype. The Dietary Approaches to Stop Hypertension(DASH) eating pattern will be prescribed to all participants in the treatment group and specific strategies to achieve goals will be discussed weekly by the participant over the phone.
  Interventions: Other: Diet and Exercise Intervention

INTERVENTIONS:
Other: Diet and Exercise Intervention — Remote Dietary and Exercise Intervention Program

SUMMARY:
The purpose of this study is to assess exercise performance in 20 healthy children 10-19 years of age with a body mass index greater than 85th percentile and to evaluate the effect of dietary and exercise intervention over 12 weeks.

DETAILED DESCRIPTION:
Our hypothesis is that the vascular health in these children will improve at the end of intervention. The results of this study will help us in our long-term objective of improving vascular health of children with congenital/acquired heart disease, a group particularly at risk for premature atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* 10-19 years old
* Overweight (BMI > 85 percentile)
* Interested in a 12 week ¬home exercise & nutrition program
* Have computer & internet access
* Can come to Lucile Packard Children's Hospital at Stanford for a 3-hour test at the start & end of the study (so only twice!)
* Are able to come to testing after fasting overnight
* Do not smoke
* Do not take any medications

Exclusion Criteria:

* non-overweight adolescents

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Vascular Health | Beginning of 12th week and end of 12th week
  Tests will include: EndoPAT analysis to assess endothelial function, applanation tonometry to assess arterial stiffness, carotid artery imaging to assess the wall thickness of the carotid arteries, exercise testing to assess the physical exercise capacity of these children and blood work to evaluate the lipid profile and inflammation status (CRP). The participant will be asked to come in after an overnight fast. They will receive a snack bag before the exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Tierney, MD, Principal Investigator — Lucile Packard Children's Hospital - Pediatric Cardiology; Chau N Vu, BS, Study Director — Lucile Packard Children's Hospital - Pediatric Cardiology; Katie Jo Buccola, Study Chair — Lucile Packard Children's Hospital - Pediatric Cardiology; Jeffrey Kazmucha, Study Chair — Lucile Packard Children's Hospital - Pediatric Cardiology; Laurie Steinberg, Study Chair — Stanford Prevention Research Center; Olga Ogareva, Study Chair — Lucile Packard Children's Hospital - Pediatric Cardiology; Inger Olson, MD, Study Chair — Lucile Packard Children's Hospital - Pediatric Cardiology; Chinyelu Nwobu, MD, Study Chair — Lucile Packard Children's Hospital - Pediatric Cardiology
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States